CLINICAL TRIAL: NCT06024655
Title: Qualitative Study to Determine How Chronic Kidney Disease is Managed by Healthcare Professionals in Primary Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 22IC7495
Record Dates: First submitted 2023-08-07; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of Chronic Kidney Disease is rising worldwide exponentially on account of a rising prevalence of the commonest causes of patients developing CKD. For instance, the prevalence of Type 2 diabetes, the commonest cause of CKD worldwide, is increasing with an expected 450 million people expected to have type 2 diabetes by 2030. Poorly controlled blood sugars are associated with a risk of complications related to the eyes, heart and kidneys amongst other organs, resulting in poor long-term health and quality of life. The kidney is one of the most frequently affected organs, with diabetes related kidney disease (DKD) the commonest cause of kidney failure worldwide, with patients requiring dialysis and transplantation to survive. However, despite transplantation allowing patients to live life's without the need for dialysis, diabetes remains to be associated with poor transplant function, cardiovascular disease and overall poor quality of life. With primary care being instrumental in the screening, diagnosis and management/monitoring of CKD, this study aims to identify areas done well as well as areas where improvement is needed to improve a patients clinical journey and management. This will be done in the form of an online questionnaire and focus groups, advertised via clinical commissioning groups across the United Kingdom. Through this, the investigators hope to gain further insight into areas of clinical management done well and areas of improvement as well as how primary care feel current management could be improved upon, obstacles faced, additional resources required and how they could be better supported by hospital specialists. Study results will be analysed and published in a peer reviewed journal with recommendations made with regards to how care should be altered to help delay and prevent CKD onset and progression.

DETAILED DESCRIPTION:
The study is designed in the form of a clinician validated online questionnaire (conducted via Qualitrics.com), with participants recruited anonymously. Integrated care boards (ICB) from across the country will be sent an online link to the questionnaire via email and encouraged to share amongst clinicians and allied health care providers within their ICB. Where participants open the study web address (via an anonymous link or QR code) they will be taken to the participant information sheet which aims to provide potential participants with more information regarding the study, its aims, benefits, risks and potential conflicts of interests. Participants will then be asked to consent to the study online following which they will be asked to complete an online questionnaire, which aims to take participants no more than fifteen minutes to complete. As an added non obligatory component, participants who complete the study, will be asked if they are willing to partake in an online focus group of uptown 6 participants in the future, to further discuss the study and gain a further understanding of factors which would empower participants to improve their individual health and diabetes control. Those participants will be asked to provide a contact email address, in order for the study organisers to make contact with the participant with regards to potential focus groups in the future. Participation is completely voluntary and participants may change their decision at any time. Participants will be consented again for their participation in the focus groups electronically prior to the focus group.Focus groups will be conducted via Microsoft Teams and will concentrate on key findings of the online questionnaire data to further understand clinician perspectives of how diabetes is currently managed and ways in which care could be improved upon. They will be of no longer than 60 minutes in duration each.

Focus groups will be audio recorded and be transcribed by the study organisers within 7 days of the focus group, following which the recording will be deleted. Transcribed focus groups will be anonymised and will be stored electronically at Imperial College London in a password protected file. Data will be analysed and submitted in the form of a research paper to a peer reviewed scientific journal.

ELIGIBILITY:
Inclusion Criteria:

Health care professional ( community based - doctor, nurse, healthcare assistant, pharmacist), working within primary care in the United Kingdom

Exclusion Criteria:

Non health care professionals Secondary care health care professionals.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Health care professional working within the primary health care system, in the United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative review of questionnaire submission and focus groups. | 6 months
  This is a qualitative study, with qualitative methods applied to analyse the data generated. The qualitative data analysis approach will systematise descriptive data collected through the online questionnaire and subsequent focus groups, with the aim being to identify patterns and themes behind the interviews, surveys, and observations and interpreting it. The method aims to identify patterns and themes behind textual data. Specific analysis undertaken will utilise: 1. Discourse analysis whereby we will review the received answers from the questionnaire and the transcript form the focus groups to determine relationships between the received information and its context. 2. Conversion of qualitative data within the online questionnaire to quantitative data to allow for conclusions to be made 3. Thematic anlaysis for the transcript of the focus group to identify themes on how patients feel their care could have been improved upon.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick W K Tam, Principal Investigator — Imperial College London; RAKESH DATTANI, Study Chair — Imperial College London; Hutan Ashrafian, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: No
No IPD data to be shared, solely aggregated data.

DOCUMENTS (1):
  • Study Protocol (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT06024655/Prot_000.pdf